CLINICAL TRIAL: NCT01544998
Title: To Define the Role of PDEV in Mediating the Decreased GFR and Attenuated Renal Sodium and cGMP Excretory Response to Acute Saline Volume Expansion in PSD and PDD With Renal Dysfunction.
Brief Title: Tadalafil and Nesiritide as Therapy in Pre-clinical Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Horng Chen, MD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 11-004257; UL1RR024150 (NIH); 5P01HL076611 (NIH)
Record Dates: First submitted 2012-01-24; First posted 2012-03-06 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tadalafil plus Placebo, then Tadalafil plus Nesiritide (Experimental): First intervention period: oral Tadalafil; after 1 hour, subcutaneous (sc) placebo given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting. There was a one week washout period. Second intervention period: oral Tadalafil; after 1 hour, sc Nesiritide given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting.
  Interventions: Drug: Nesiritide; Drug: Tadalafil; Drug: Placebo; Drug: Saline load
- Tadalafil plus Nesiritide, then Tadalafil plus Placebo (Experimental): First intervention period: oral Tadalafil; after 1 hour, sc Nesiritide given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting. There was a one week washout period. Second intervention period: oral Tadalafil; after 1 hour, sc placebo given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting.
  Interventions: Drug: Nesiritide; Drug: Tadalafil; Drug: Placebo; Drug: Saline load

INTERVENTIONS:
Drug: Nesiritide — 10 ug/kg
Drug: Tadalafil — 5 mg
  Other Names: Cialis; Adcira
Drug: Placebo — The pharmacy will create a placebo subcutaneous injection volume to match the volume of Nesiritide dose.
Drug: Saline load — Normal saline 0.9% 0.25 ml/kg/min for 60 minutes

SUMMARY:
This study is being done to determine the effects of subcutaneous (under the skin) injection of human B-type natriuretic factor (BNP), Natrecor (nesiritide), a hormone produced by the heart, in combination with Tadalafil on:

* The pumping function of the heart
* Kidney function
* Hormonal function (levels of different hormones in your blood) in persons with lower pumping function of their heart.

DETAILED DESCRIPTION:
In the American Heart Association/American College of Cardiology classification of heart failure (HF), stage B is defined as patients with abnormal heart structure/function (systolic or diastolic dysfunction) without symptoms. This concept of preclinical HF is based on the fact that abnormal heart structure/function can be detected by complementary methods before the development of symptoms. Patients with those abnormalities may progress to heart failure and are at increased risk of adverse cardiac events. Preclinical systolic dysfunction (PSD) is the initial compensated phase of left ventricular systolic dysfunction without symptoms of HF. We have established that diastolic dysfunction is common in the general population being present in approximately 25% of the population over age 45, the majority of whom are asymptomatic i.e., preclinical diastolic dysfunction (PDD). Cyclic guanosine monophosphate (cGMP) is the second messenger of the natriuretic peptide system (NPS) and the nitric oxide system (NO) and plays an important role in the preservation of myocardial, vascular, and renal function. Hence, disruption of this signal transduction process may contribute to the development of cardiorenal dysfunction. Type V phosphodiesterase (PDEV) metabolizes cGMP and is abundant in the kidney, vasculature, and has been recently reported in the heart. We and others have demonstrated that renal PDEV is up-regulated in experimental HF and may lead to the attenuation of renal cGMP generation in response to both endogenous and exogenous BNP, thus serving as a mechanism for renal resistance to BNP. Furthermore, in experimental overt HF, 10 days of PDEV inhibition treatment resulted in reduction of left ventricular (LV) mass, increased LV fractional shortening and cardiac output but did not improve renal function. However, chronic PDEV inhibition did enhance the renal actions of exogenous BNP, specifically improving glomerular filtration rate (GFR) and renal cGMP generation. PDEV inhibitors are FDA approved for erectile dysfunction and pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (PSD)

* an ejection fraction of less than 45% with no clinical signs or symptoms of congestive heart failure;
* a minimal distance on 6-minute walk of >450 meters
* calculated creatinine clearance of equal or less than 90 ml/min and greater than 30 ml/min, using the Modification of Diet in Renal Disease (MDRD) formula assessed within the past 24 months. If the creatinine clearance is > 24 months a creatinine test can be drawn at screen/enrollment visit.
* A 6-minute walk distance of 450 meters

Group 2 (PDD)

* ejection fraction of greater than 50% with moderate or severe diastolic dysfunction as assessed by Doppler echocardiography,
* who do not have any signs or symptoms of congestive heart failure
* minimal distance on 6-minute walk of >450 meters
* calculated creatinine clearance of equal or less than 90 ml/min and greater than 30 ml/min

Exclusion Criteria:

* Current or anticipated future need for nitrate therapy
* Systolic blood pressure < 90 mmHg or > 180 mm Hg
* Diastolic blood pressure < 40 mmHg or > 100 mmHg
* Resting heart rate (HR) > 100 bpm
* Patients taking alpha antagonists or cytochrome P450 3A4 inhibitors (ketoconazole, itraconazole, erythromycin, saquinavir, cimetidine or serum protease inhibitors for HIV).
* Patients with retinitis pigmentosa, previous diagnosis of nonischemic optic neuropathy, untreated proliferative retinopathy or unexplained visual disturbance
* Patients with sickle cell anemia, multiple myeloma, leukemia or penile deformities placing them at risk for priapism (angulation, cavernosal fibrosis or Peyronie's disease)
* Contraindication to nesiritide.
* Patients with an allergy to iodine.
* Valve disease (> moderate aortic or mitral stenosis; > moderate aortic or mitral regurgitation)
* Hypertrophic cardiomyopathy
* Infiltrative or inflammatory myocardial disease (amyloid, sarcoid)
* Pericardial disease
* Have experienced a myocardial infarction or unstable angina, or have undergone percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) within 60 days prior to consent, or requires either PTCA or CABG at the time of consent
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening or other evidence of significantly compromised central nervous system (CNS) perfusion
* Patients with severe liver disease (AST > 3x normal, alkaline or bilirubin > 2x normal)
* Serum sodium of < 125 milliequivalents (mEq)/dL or > 150 mEq/dL
* Serum potassium of < 3.2 mEq/dL or > 5.7 mEq/dL
* Prior diagnosis of intrinsic renal diseases including renal artery stenosis of > 50%
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Less than 21 years of age
* Pregnant or nursing women.
* Women of child bearing potential who do not have a negative pregnancy test at study entry and who are not using effective contraception

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H Chen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wan SH, McKie PM, Slusser JP, Burnett JC Jr, Hodge DO, Chen HH. Effects of phosphodiesterase V inhibition alone and in combination with BNP on cardiovascular and renal response to volume load in human preclinical diastolic dysfunction. Physiol Rep. 2021 Aug;9(16):e14974. doi: 10.14814/phy2.14974. PMID 34405565
- [Derived] Wan SH, Torres-Courchoud I, McKie PM, Slusser JP, Redfield MM, Burnett JC Jr, Hodge DO, Chen HH. Cardiac Versus Renal Response to Volume Expansion in Preclinical Systolic Dysfunction With PDEV Inhibition and BNP. JACC Basic Transl Sci. 2019 Dec 23;4(8):962-972. doi: 10.1016/j.jacbts.2019.08.008. eCollection 2019 Dec. PMID 31909303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 2 participants in the Preclinical Systolic Dysfunction group withdrew from the study before they were randomized. No participant in the Preclinical Diastolic Dysfunction group withdrew.
Period: First Intervention (3 Hours)
Arm/Group | Tadalafil Plus Placebo, Then Tadalafil Plus Nesiritide | Tadalafil Plus Nesiritide, Then Tadalafil Plus Placebo
Started | 26 | 15
Completed | 26 | 15
Not Completed | 0 | 0
Period: Washout (1 Week)
Arm/Group | Tadalafil Plus Placebo, Then Tadalafil Plus Nesiritide | Tadalafil Plus Nesiritide, Then Tadalafil Plus Placebo
Started | 26 | 15
Completed | 26 | 15
Not Completed | 0 | 0
Period: Second Intervention (3 Hours)
Arm/Group | Tadalafil Plus Placebo, Then Tadalafil Plus Nesiritide | Tadalafil Plus Nesiritide, Then Tadalafil Plus Placebo
Started | 26 | 15
Completed | 26 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population description includes only those subjects who completed the study.
Groups:
- Entire Study Population: Includes groups randomized to receive Tadalafil plus Nesiritide first, and Tadalafil plus Placebo first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Natriuresis (Urinary Sodium Excretion) at 60 Minutes for Preclinical Systolic Dysfunction (PSD) Reporting Group
Description: Value at 60 minutes minus value at baseline.
Time Frame: Baseline, 60 minutes after saline load
Population: This was a within PSD reporting group comparison; between PSD and PDD groups were not compared.
Measure: Mean (Standard Deviation); unit: mEq/min
Groups:
- Tadalafil Plus Nesiritide: Oral Tadalafil; after 1 hour, sc Nesiritide given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting. This dosing administration was in either first intervention period or second intervention period.
- Tadalafil Plus Placebo: Oral Tadalafil; after 1 hour, subcutaneous (sc) placebo given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting. This dosing administration was in either first intervention period or second intervention period.
Arm/Group | Tadalafil Plus Nesiritide | Tadalafil Plus Placebo
Number analyzed (Participants) | 21 | 21
mEq/min | 41.8 (161.8) | 88.9 (86.5)
Statistical Analysis 1: Comparison: Tadalafil Plus Nesiritide vs Tadalafil Plus Placebo; This was a within PSD reporting group comparison; between PSD and PDD groups were not compared; Test type: Superiority or Other; p = 0.26, t-test, 2 sided

2. Primary Outcome: Change in Natriuresis (Urinary Sodium Excretion) at 60 Minutes for Preclinical Diastolic Dysfunction (PDD) Reporting Group
Description: Value at 60 minutes minus value at baseline.
Time Frame: Baseline, 60 minutes after saline load
Population: This was a within PDD reporting group comparison; between PSD and PDD groups were not compared.
Measure: Mean (Standard Deviation); unit: mEq/min
Arm/Group | Tadalafil Plus Nesiritide | Tadalafil Plus Placebo
Number analyzed (Participants) | 20 | 20
mEq/min | 92.5 (185) | 97.0 (183)
Statistical Analysis 1: Comparison: Tadalafil Plus Nesiritide vs Tadalafil Plus Placebo; This was a within PDD reporting group comparison; between PSD and PDD groups were not compared; Test type: Superiority or Other; p = 0.90, t-test, 2 sided

3. Secondary Outcome: Change in Glomerular Filtration Rate (GFR) at 60 Minutes for Preclinical Systolic Dysfunction (PSD) Reporting Group
Description: Value at 60 minutes minus value at baseline.
Time Frame: Baseline, 60 minutes after saline load
Population: This was a within PSD reporting group comparison; between PSD and PDD groups were not compared.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Tadalafil Plus Nesiritide | Tadalafil Plus Placebo
Number analyzed (Participants) | 21 | 21
mL/min/1.73 m^2 | -12.7 (21.2) | 9.4 (22.7)
Statistical Analysis 1: Comparison: Tadalafil Plus Nesiritide vs Tadalafil Plus Placebo; This was a within PSD reporting group comparison; between PSD and PDD groups were not compared; Test type: Superiority; p = 0.003, t-test, 2 sided

4. Secondary Outcome: Change in Glomerular Filtration Rate (GFR) at 60 Minutes for Preclinical Diastolic Dysfunction (PDD) Reporting Group
Description: Value at 60 minutes minus value at baseline.
Time Frame: Baseline, 60 minutes after saline load
Population: This was a within PDD reporting group comparison; between PSD and PDD groups were not compared.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Tadalafil Plus Nesiritide | Tadalafil Plus Placebo
Number analyzed (Participants) | 20 | 20
mL/min/1.73 m^2 | -5.3 (26.1) | 3.9 (24.3)
Statistical Analysis 1: Comparison: Tadalafil Plus Nesiritide vs Tadalafil Plus Placebo; This was a within PDD reporting group comparison; between PSD and PDD groups were not compared; Test type: Superiority; p = 0.14, t-test, 2 sided

5. Secondary Outcome: Change in Urinary Cyclic Guanosine Monophosphate (cGMP) at 60 Minutes for Preclinical Systolic Dysfunction (PSD) Reporting Group
Description: Value at 60 minutes minus value at baseline.
Time Frame: Baseline, 60 minutes after saline load
Population: This was a within PSD reporting group comparison; between PSD and PDD groups were not compared.
Measure: Mean (Standard Deviation); unit: pmol/min
Arm/Group | Tadalafil Plus Nesiritide | Tadalafil Plus Placebo
Number analyzed (Participants) | 20 | 20
pmol/min | 2566.9 (1888.3) | 34.2 (354.9)
Statistical Analysis 1: Comparison: Tadalafil Plus Nesiritide vs Tadalafil Plus Placebo; This was a within PSD reporting group comparison; between PSD and PDD groups were not compared; Test type: Superiority; p < 0.001, t-test, 2 sided

6. Secondary Outcome: Change in Urinary Cyclic Guanosine Monophosphate (cGMP) at 60 Minutes for Preclinical Diastolic Dysfunction (PDD) Reporting Group
Description: Value at 60 minutes minus value at baseline.
Time Frame: Baseline, 60 minutes after saline load
Population: This was a within PSD reporting group comparison; between PSD and PDD groups were not compared.
Measure: Mean (Standard Deviation); unit: pmol/min
Arm/Group | Tadalafil Plus Nesiritide | Tadalafil Plus Placebo
Number analyzed (Participants) | 20 | 20
pmol/min | 1851 (1386.4) | 173.4 (517.9)
Statistical Analysis 1: Comparison: Tadalafil Plus Nesiritide vs Tadalafil Plus Placebo; This was a within PDD reporting group comparison; between PSD and PDD groups were not compared; Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through 7 days after the completion of the second study day.
Groups:
- PSD: Tadalafil Plus Nesiritide; PDD: Tadalafil Plus Nesiritide: Oral Tadalafil; after 1 hour, sc Nesiritide given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting. This dosing administration was in either first intervention period or second intervention period.
- PSD: Tadalafil Plus Placebo; PDD: Tadalafil Plus Placebo: Oral Tadalafil; after 1 hour, subcutaneous (sc) placebo given in the abdomen. After a lead in period of 15 min, a 30-min clearance was repeated, then acute saline load was given. During the 1 hour saline load, one 30-min clearance repeated with subject in supine position, then second 30-min clearance repeated with subject sitting. This dosing administration was in either first intervention period or second intervention period.
Arm/Group | PSD: Tadalafil Plus Nesiritide | PSD: Tadalafil Plus Placebo | PDD: Tadalafil Plus Nesiritide | PDD: Tadalafil Plus Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/21 | 0/21 | 4/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PSD: Tadalafil Plus Nesiritide (N=21) | PSD: Tadalafil Plus Placebo (N=21) | PDD: Tadalafil Plus Nesiritide (N=20) | PDD: Tadalafil Plus Placebo (N=20)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IV Site Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes